CLINICAL TRIAL: NCT00262327
Title: Phase I Trial of Intratumoral Injection of an Adenovirus Encoding Human Endostatin for Advanced Solid Tumors
Brief Title: Safety and Efficacy of Adenoviral Endostatin in the Treatment of Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Doublle Bioproduct Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DB-101; E10A
Record Dates: First submitted 2005-12-02; First posted 2005-12-06 (Estimated); Last update posted 2006-06-20 (Estimated); Status verified 2005-12

CONDITIONS: Advanced Solid Tumor
Keywords: antiangiogenesis; endostatin; adenovirus; gene therapy; cancer
MeSH Terms: conditions — Adenoviridae Infections; Neoplasms | interventions — Endostatins

INTERVENTIONS:
Drug: Antangiogenesis
Genetic: endostatin gene

SUMMARY:
The growth and metastasis of solid tumors are dependent on angiogenesis. Endostatin, the C-terminal proteolytic fragment of collagen XVIII, is an effective endogenous angiogenesis inhibitor in cancer therapy in mice. Applied for clinical studies in solid tumor, however, recombinant human endostatin protein, difficulties in a large-scale production of the recombinant endostatin protein, and the cumbersome daily administration. Up to now, its clinical application has been hampered by those matters. We herein constructed a adenoviral vector ecoding human endostatin. This study will test the safety and efficacy of recombinant human endostatin adenovirus (Ad-rhE) in the treatment of patients with advanced solid tumors.

DETAILED DESCRIPTION:
It is widely recognized that angiogenesis not only is important in physiological processes such as embryonic development, wound healing, and organ and tissue regeneration, but also play a pivotal role in tumor growth, tissue invasion, and metastasis.1 This complex, multistep process of angiogenesis involves interactions between tumor cells and endothelial cells (ECs), growth factors, and extracellular matrix components. Tumors that are unable to elicit angiogenesis exist in a dormant state, and are unable to grow beyond the size of 1-2 mm. Angiogenesis is regulated by a variety of pro-angiogenesis and anti-angiogenesis factors and their imbalance can lead to disease. The abnormal features of the tumor vasculature perhaps represent an imbalanced expression of proangiogenic factors and antiangiogenic factors.1 Antiangiogenic therapies inhibit the growth of genetically stable endothelial cells, and most tumors should starve to death with little acquired resistance. Antiangiogenesis agents such as Avastin for the treatment of cancer have now been approved by the FDA in the US and in other countries.2 Endostatin, a 20 kDa C-terminal fragment of the carboxyterminus of collagen XVIII, has been shown to block endothelial cell proliferation, survival, and migration, in part through downregulating proangiogenic factor (such as Ids, HIF-1a, VEGF-A, bFGF) and upregulating antiangiogenic factors (such as Thrombospondin-1,2, vasostatin, kininogen).4,5,6 Of the endogenous antiangiogenic factors in the body, endostatin has broadest anti-cancer spectrum and the least toxic and no resistance anti-cancer drug in mice and human. Endostatin is the first endogenous angiogenesis inhibitor to introduce into human clinical trials.

However, therapy with recombinant endostatin protein is hampered by their shot half-life, difficulties in protein production and long-term storage of bioactive protein. Furthermore, the inhibition of tumor angiogenesis is a long-term and chronic process of treatment. Gene therapy may be overcome these difficulties by introducing human endostatin cDNA into the host and using the body as an endogenous factory to generate highly bioactive gene product. Expression of endostatin by adenoviral gene transfer (Ad-rhEndo, E10A) generates a strong systemic therapeutic effect in several models of solid tumors in mice.7,8,9,10 Intratumoral injections of E10A into subcutaneous xenografts of hepatocellular carcinoma BEL-7402, nasopharyngeal carcinoma CNE-2, Tongue cancer Tca8113 in nude mice demonstrated significant tumor growth inhibition and reduce angiogenesis in tumors. No toxic effects of E10A administration in these pharmacology studies were identified. On the base of promising preclinical results in solid tumors, we undertook a dose-escalation phase I trial of E10A in the treatment of patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years;
* Genders eligible for study: both;
* Histologic diagnosis of solid malignancies ;
* Performance status of 0 or 1;
* Tumor not amenable to standard curative or palliative therapy;
* An accessible tumor mass;
* At least 4 weeks since prior biotherapy/chemotherapy/radiotherapy;
* A life expectancy beyond 3 months;
* Ability to give signed informed consent.

Exclusion Criteria:

* Pregnancy or lactation;
* Had a history of brain metastasis or a primary brain tumor;
* An active, potentially severe autoimmune disease;
* Serum creatinine ≥1.5mg/dl or a calculated creatinine clearance <60ml/min;
* WBC count < 2.0×109/L，hemoglobin < 90g/L，and platelet count < 100×109/L;
* Total bilirubin value < 2.0 times the upper limit of normal (ULN), ALT level < 2.0 times ULN, AST < 2.0 times ULN;
* Positive of anti-HIV antibodies;
* An active bacterial, fungal, or viral infection;
* Less than one month since prior systemic immunosuppressive drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-05; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Overall Officials: Wenqi Jiang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China